CLINICAL TRIAL: NCT04799054
Title: Phase 1/2, Open-label, Dose Escalation and Dose Expansion Study of TransCon TLR7/8 Agonist Alone or in Combination With Pembrolizumab in Participants With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Study of TransCon TLR7/8 Agonist With or Without Pembrolizumab in Patients With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor made the decision to close enrollment to prioritize our efforts on TransCon IL-2 ß/g.
Sponsor: Ascendis Pharma Oncology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCTLR-101; transcendIT-101 (Other: Ascendis Pharma)
Record Dates: First submitted 2021-02-26; First posted 2021-03-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Locally Advanced Solid Tumor; Metastatic Solid Tumor; Head and Neck Squamous Cell Carcinoma HNSCC; HPV-associated Cancers; Neoadjuvant Melanoma; Neoadjuvant Cutaneous Squamous Cell Carcinoma (cSCC)
Keywords: Ascendis Pharma; TransCon TLR7/8 Agonist; Locally Advanced Solid Tumor; Metastatic Solid Tumor; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Monotherapy Dose Escalation and Optimization: TransCon TLR7/8 Agonist (Experimental): TransCon TLR7/8 Agonist in escalating doses to evaluate safety/tolerability and to determine the MTD and RP2D.
  Interventions: Drug: TransCon TLR7/8 Agonist
- Part 2 Combination Dose Escalation and Optimization: TransCon TLR7/8 Agonist with Pembrolizumab (Experimental): TransCon TLR7/8 Agonist with Pembrolizumab in escalating doses to evaluate safety/tolerability and determine the MTD and RP2D.
  Interventions: Drug: TransCon TLR7/8 Agonist; Drug: Pembrolizumab
- Part 3 Phase 2 Combination Dose Expansion: TransCon TLR7/8 Agonist with Pembrolizumab (Experimental): TransCon TLR7/8 Agonist with Pembrolizumab using RP2D from Part 2 to evaluate safety/tolerability and anti-tumor activity of the combination in indication-specific dose expansion cohorts.
  Interventions: Drug: TransCon TLR7/8 Agonist; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TransCon TLR7/8 Agonist — TransCon TLR7/8 Agonist will be administered as an IT injection
Drug: Pembrolizumab — Pembrolizumab will be administered IV
  Arms: Part 2 Combination Dose Escalation and Optimization: TransCon TLR7/8 Agonist with Pembrolizumab; Part 3 Phase 2 Combination Dose Expansion: TransCon TLR7/8 Agonist with Pembrolizumab

SUMMARY:
TransCon TLR7/8 Agonist is an investigational drug being developed for treatment of locally advanced or metastatic solid tumors. This Phase 1/2 study will evaluate TransCon TLR7/8 Agonist as monotherapy or in combination with pembrolizumab in dose escalation and dose expansion. Participants will receive intratumoral (IT) injection of TransCon TLR7/8 Agonist every cycle. The primary objectives are to evaluate safety and tolerability, and define the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab.

DETAILED DESCRIPTION:
Toll-like receptors (TLRs) are a class of proteins that play a key role in innate immune cell recognition of foreign pathogens, stimulating innate and adaptive immune responses. TransCon TLR7/8 Agonist is designed as a long-acting localized delivery prodrug of resiquimod, a potent toll-like receptor (TLR) 7/8 agonist, with the potential to prolong high local concentrations of resiquimod and promote potent anti-tumoral responses while reducing systemic drug exposure and related adverse events. TransCon TLR7/8 Agonist is expected to stimulate innate and adaptive immune response in the tumor microenvironment and enhance the activity of checkpoint inhibitors like pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Participants must have histologically confirmed locally advanced, recurrent or metastatic solid tumor malignancies that cannot be treated with curative intent (surgery or radiotherapy).
* Participants must have progressed on or be intolerant of available standard of care treatment options or have disease for which there is no standard of care treatment available, with the exception of participants enrolling to the neoadjuvant cohorts.
* At least 2 lesions of measurable disease, unless specified otherwise in the selection criteria.
* Willingness to undergo biopsies.
* Demonstrated adequate organ function within 28 days of Cycle 1 Day 1 (C1D1).
* Life expectancy >12 weeks as determined by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Participants who have undergone treatment with anti-PD-1, anti-PD-L1, or antiCTLA 4 antibody must have at least 4 weeks from the last dose of antibody and evidence of disease progression per investigator assessment before enrollment.
* Participants who have previously received an immune checkpoint inhibitor prior to enrollment must have any immune related toxicities resolved to ≤Grade 1 or baseline (prior to the checkpoint inhibitor) to be eligible.
* Female and male participants of childbearing potential who are sexually active must agree to use highly effective methods of contraception.

Exclusion Criteria:

* Participants who have been previously treated with a TLR agonist (excluding topical agents for unrelated disease) are not eligible.
* Other active malignancies within the last 2 years are excluded.
* Active autoimmune diseases, regardless of need for immunosuppressive treatment at the time of screening, with the exception of patients well controlled on physiologic endocrine replacement.
* Systemic immunosuppressive treatment with the exception for patients on corticosteroid taper (for example, for chronic obstructive pulmonary disease exacerbation). Participants cannot start dosing on study until steroid dose is at or lower than 10 mg per day prednisone or equivalent.
* Women who are breastfeeding or have a positive serum pregnancy test during screening or within 72 hours prior to C1D1 are not eligible.
* Vaccination with live, attenuated vaccines within 4 weeks of enrollment.
* Symptomatic central nervous system metastases.
* Known bleeding disorder that is deemed to place the patient at unacceptable risk for bleeding complications from intratumoral injections or biopsies.
* Known hypersensitivity to any component of TransCon TLR7/8 Agonist or pembrolizumab.
* Any uncontrolled bacterial, fungal, viral, or other infection.
* Treatment with any other anti-cancer systemic treatment (approved or investigational) or radiation therapy within 4 weeks of first dosing on study is not allowed.
* Significant cardiac disease
* A marked baseline prolongation of QT/QTc (corrected QT) interval (e.g., repeated demonstration of a QTc interval >480 ms (National Cancer Institute NCI) Common Terminology Criteria for Adverse Events [CTCAE] grade 1) using Fredericia's QT correction formula.
* A history of additional risk factors for Torsades de Pointes (TdP) (e.g., heart failure, clinically significant hypokalemia, family history of Long QT Syndrome).
* The use of concomitant medications that prolong the QT/QTc interval within 14 days of enrollment.
* Positive for HIV or with active hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, expected average of 2 years
  Treatment emergent and treatment related adverse events (assessed by CTCAE v5.0), serious adverse events (SAEs), adverse events leading to treatment discontinuation, deaths
Maximum Tolerated Dose (MTD) | Cycle 1 (each cycle is 21 days) in Part 1 (monotherapy dose escalation) and Cycle 1 (the first cycle is 28 days and 21 days thereafter) in Part 2 (combination therapy dose escalation)
  Determine the maximum tolerated dose by assessing the Incidence of Dose Limiting Toxicities (DLTs), treatment emergent and treatment related adverse events (assessed by CTCAE v5.0), serious adverse events (SAEs), adverse events leading to treatment discontinuation and deaths.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of TransCon TLR7/8 Agonist and combination regimen for further development by evaluating number of patients with treatment-related adverse events as assessed by CTCAE.
Response | 9 weeks
  Evaluate the Pathologic complete response (pCR) per local assessment for pathology review anti-tumor activity of TransCon TLR7/8 Agonist in combination with pembrolizumab in the Neoadjuvant Cohorts

SECONDARY OUTCOMES:
Overall Response Rate | Average of two years
  Response assessed by RECIST v1.1 and itRECIST (response assessment for intratumoral immunotherapy for injected and noninjected lesions)
Duration of Response | Average of two years
  Time from first documentation of objective tumor response (CR or PR that is subsequently confirmed) to first documentation of disease progression or death due to any cause, whichever occurs first
Time to Response | Expected up to 1 year from first dose
  Time from date of first dose of study treatment to first occurrence of response (CR or PR)
Progression Free Survival (PFS) | Average of two years
  Time from date of first dose of study treatment to first documentation of disease progression or death due to any cause
Event free survival (EFS) by RECIST 1.1 per investigator assessment | Average of two years
Overall Survival (OS) | Average of two years
  Time from date of first dose of study treatment to date of death due to any cause
PK characterization - Cmax | Average of two years
  Maximum observed plasma concentration of resiquimod, O-desethyl resiquimod (metabolite) and total resiquimod (sum of bound and unbound resiquimod) after IT administration of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab
PK characterization - tmax | Average of two years
  Time to reach maximum plasma concentration of resiquimod, O-desethyl resiquimod (metabolite) and total resiquimod (sum of bound and unbound resiquimod) after IT administration of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab
PK characterization - AUC0-t for first dose only | Average of two years
  Area under the plasma concentration-time curve from time zero to last sampling time at which the concentration is at or above the lower limit of quantification for resiquimod, O-desethyl resiquimod (metabolite) and total resiquimod (sum of bound and unbound resiquimod) after IT administration of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab
PK characterization - t1/2 | Average of two years
  Apparent terminal half-life of resiquimod, O-desethyl resiquimod (metabolite) and total resiquimod (sum of bound and unbound resiquimod) after IT administration of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab
PK characterization - Ctrough | Average of two years
  Plasma concentration immediately before next dosing of resiquimod, O-desethyl resiquimod (metabolite) and total resiquimod (sum of bound and unbound resiquimod) after IT administration of TransCon TLR7/8 Agonist alone or in combination with pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Joan Morris, Study Director — Medical Monitor
Locations (37):
- United States (16):
  - Ascendis Pharma Investigational Site, Duarte, California
  - Ascendis Investigational Site, Los Angeles, California
  - Ascendis Investigational Site, Orange, California
  - Ascendis Pharma Investigational Site, San Francisco, California
  - Ascendis Investigational Site, Tampa, Florida
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Iowa City, Iowa
  - Ascendis Pharma Investigational Site, Louisville, Kentucky
  - Ascendis Pharma Investigational Site, Canton, Ohio
  - Ascendis Pharma Investigational Site, Cincinnati, Ohio
  - Ascendis Pharma Investigational Site, Cleveland, Ohio
  - Ascendis Pharma Investigational Site, Pittsburgh, Pennsylvania
  - Ascendis Pharma Investigational Site, Knoxville, Tennessee
  - Ascendis Investigational Site, Dallas, Texas
  - Ascendis Investigational Site, Houston, Texas
  - Ascendis Pharma Investigational Site, Fairfax, Virginia
- Australia (3):
  - Ascendis Pharma Investigational Site, Wollongong, New South Wales
  - Ascendis Pharma Investigational Site, Frankston, Victoria
  - Ascendis Investigational Site, Bedford Park
- Netherlands (2):
  - Ascendis Investigational Site, Amsterdam
  - Ascendis Investigational Site, Rotterdam
- South Korea (6):
  - Ascendis Investigational Site, Dalseo-gu
  - Ascendis Investigational Site, Seocho-gu
  - Ascendis Investigational Site, Seogu
  - Ascendis Investigational Site, Seongnam
  - Ascendis Investigational Site, Seoul
  - Ascendis Investigational Site, Suwon
- Spain (7):
  - Ascendis Investigational Site, Barcelona
  - Ascendis Investigational Site, Madrid
  - Ascendis Investigational Site, Málaga
  - Ascendis Investigational Site, Murcia
  - Ascendis Investigational Site, Pamplona
  - Ascendis Investigational Site, Seville
  - Ascendis Investigational Site, Valencia
- Taiwan (3):
  - Ascendis Investigational Site, Taichung
  - Ascendis Investigational Site, Tainan
  - Ascendis Investigational Site, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lessmann T, Jones SA, Voigt T, Weisbrod S, Kracker O, Winter S, Zuniga LA, Stark S, Bisek N, Sprogoe K. Degradable Hydrogel for Sustained Localized Delivery of Anti-Tumor Drugs. J Pharm Sci. 2023 Nov;112(11):2843-2852. doi: 10.1016/j.xphs.2023.05.018. Epub 2023 Jun 4. PMID 37279836
- [Derived] Zuniga LA, Lessmann T, Uppal K, Bisek N, Hong E, Rasmussen CE, Karlsson JJ, Zettler J, Holten-Andersen L, Bang K, Thakar D, Lee YC, Martinez S, Sabharwal SS, Stark S, Faltinger F, Kracker O, Weisbrod S, Muller R, Voigt T, Bigott K, Tabrizifard M, Breinholt VM, Mirza AM, Rosen DB, Sprogoe K, Punnonen J. Intratumoral delivery of TransCon TLR7/8 Agonist promotes sustained anti-tumor activity and local immune cell activation while minimizing systemic cytokine induction. Cancer Cell Int. 2022 Sep 19;22(1):286. doi: 10.1186/s12935-022-02708-6. PMID 36123697